CLINICAL TRIAL: NCT03009097
Title: "Comparative Evaluation Of The Efficacy Of Atorvastatin Gel As An Adjunct To Allografts In The Treatment Of Intrabony Defects" - A Clinico Radiological Study
Brief Title: Atorvastatin as an Adjunct to DFDBA in Intrabony Defects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kamineni Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, ETIKA RATHI, Principal investigator, Kamineni Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kamineni perio
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Periaortitis; Intrabony Periodontal Defect
Keywords: Chronic periodontitis; atorvastatin; intrabony defect
MeSH Terms: conditions — Retroperitoneal Fibrosis; Chronic Periodontitis | interventions — Transplantation, Homologous; Atorvastatin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- DFDBA (Active Comparator): 13 intrabony defects in chronic periodontitis patients were treated with DFDBA
  Interventions: Biological: DFDBA
- DFDBA with Atorvastatin (Active Comparator): 13 intrabony defects in chronic periodontitis patients were treated with DFDBA in combination with Atorvastatin gel.
  Interventions: Drug: DFDBA with atorvastatin

INTERVENTIONS:
Biological: DFDBA — 13 intrabony defects in chronic periodontitis patients were treated with allograft (DFDBA)
  Other Names: Allograft
  Arms: DFDBA
Drug: DFDBA with atorvastatin — 13 intrabony defects in chronic periodontitis patients were treated with allograft (DFDBA) in combination with atorvastatin gel
  Other Names: atorvastatin gel
  Arms: DFDBA with Atorvastatin

SUMMARY:
Periodontitis is a major oral health problem which leads to the progressive destruction of periodontal ligament and alveolar bone with pocket formation, recession or both. The ultimate goal of periodontal therapy is to regenerate the lost periodontal tissue. The most common form of regenerative periodontal therapy is the use of bone grafts which stimulate bone formation by the processes of osteoinduction and osteoconduction.

Statins are a group of lipid lowering drugs which inhibit bone resorption by inhibition of the enzyme HMG-CoA reductase. They also stimulate new bone formation by local stimulation of BMP-2, a major bone growth regulatory factor. They also have anti-inflammatory and anti oxidant properties.

Very few studies exist evaluating the beneficiary effects of grafts if combined with the statins which might enhance the regeneration by bone grafts.

Hence, the present study was carried out in an attempt to comparatively evaluate clinically and radiologically, the efficacy of atorvastatin gel as an adjunct to allograft in the treatment of intrabony defects.

DETAILED DESCRIPTION:
A total of 26 intrabony defects in patients with chronic periodontitis as diagnosed by radiographs, were selected for the study after taking an informed consent. The selected sites were randomized in 2 treatment groups.

Group I - sites were treated with allograft (DFDBA) Group II - sites were treated with allograft (DFDBA) in combination with Atorvastatin gel.

Clinical parameters like probing depth and clinical attachment level and radiological assessment of intrabony defect fill were done at baseline and 3 and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy individual based on personal and medical history.
2. Presentation of untreated Chronic Periodontitis with intrabony defect having probing pocket depth (PPD) ≥5mm or clinical attachment loss of ≥ 3mm and radiographic signs of angular bone loss.

Exclusion Criteria:

1. Patients diagnosed and treated for systemic disease
2. Pregnant and Lactating women
3. Smokers
4. History of allergy to statin group or patients on systemic statin therapy.
5. History of antibiotic or periodontal therapy for the past 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
bone fill in mm was measured by taking radiographs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Etika Rathi, MDS, Principal Investigator — Kamineni Institute of Dental Sciences

REFERENCES:
- [Background] Pradeep AR, Kumari M, Rao NS, Martande SS, Naik SB. Clinical efficacy of subgingivally delivered 1.2% atorvastatin in chronic periodontitis: a randomized controlled clinical trial. J Periodontol. 2013 Jul;84(7):871-9. doi: 10.1902/jop.2012.120393. Epub 2012 Oct 2. PMID 23030241